CLINICAL TRIAL: NCT02163733
Title: An Open-label, Randomised, Phase I, Study to Determine the Effect of Food on the Pharmacokinetics of Single Oral Doses of AZD9291 in Patients With EGFRm Positive NSCLC Whose Disease Has Progressed on an EGFR TKI
Brief Title: Study to Determine the Effect of Food on the Blood Levels of AZD9291 Following Oral Dosing of a Tablet Formulation in Patients With Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Masking: None | Purpose: Other
Other Study IDs: D5160C00009; 2014-001556-37 (EudraCT Number)
Record Dates: First submitted 2014-05-29; First posted 2014-06-16 (Estimated); Results first posted 2016-04-05 (Estimated); Last update posted 2024-01-22 (Actual); Status verified 2023-12

CONDITIONS: Advanced Non Small Cell Lung Cancer; Advanced (Inoperable) Non Small Cell Lung Cancer
Keywords: oncology, cancer, non small cell lung cancer, anticancer drug, pharmacokinetics, AZD9291, EGFR sensitivity mutation, food effect
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Neoplasms | interventions — osimertinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fasted (Other): AZD9291 tablets following a period of fasting
  Interventions: Drug: AZD9291 tablets; Procedure: Pharmacokinetic sampling - AZD9291; Other: Dietary Fasted; Procedure: Pharmacokinetic sampling - AZ5140 and AZ7550
- High-fat meal (Other): AZD9291 tablets following a high-fat meal.
  Interventions: Drug: AZD9291 tablets; Procedure: Pharmacokinetic sampling - AZD9291; Other: Dietary High Fat; Procedure: Pharmacokinetic sampling - AZ5140 and AZ7550

INTERVENTIONS:
Drug: AZD9291 tablets — AZD9291 tablets: Part A 80mg od, days 1 and 10 only. Part B 80mg od for 12 months.
Procedure: Pharmacokinetic sampling - AZD9291 — Blood samples taken pre and post dosing of AZD9291 following either a period of fasting or consumption of a meal.
Other: Dietary Fasted — Fasted from 10 hours prior to dosing with 80mg AZD9291 tablet and 4 hours after dosing
  Arms: Fasted
Other: Dietary High Fat — Allocated breakfast prior to dosing with 80mg AZD9291 tablet
  Arms: High-fat meal
Procedure: Pharmacokinetic sampling - AZ5140 and AZ7550 — Blood samples taken pre and post dosing of AZD9291 following either a period of fasting or consumption of a meal.

SUMMARY:
This is a 2-part study in patients with epidermal growth factor receptor mutation positive (EGFRm+) non-small cell lung cancer (NSCLC) whose disease has progressed on treatment with an epidermal growth factor receptor (EGFR)-tyrosine kinase inhibitor (TKI): Part A will determine the effect of food on the pharmacokinetics (PK) of AZD9291; Part B will allow patients further access to AZD9291 and will provide for additional safety data collection.

Part A is a randomised, open-label, 2 treatment period crossover study in which patients will each receive a single oral dose of AZD9291 (1 x 80 mg tablet) at breakfast time (approximately 0800) in each of 2 treatment periods (once immediately following a high fat meal [fed], and once in the fasted state [fasted]), with a washout period of 9 days between doses.

Approximately 38 patients are planned to be enrolled and dosed; at least 30 evaluable patients will be required to complete Part A (ie, the last PK sample in Treatment Period 2 [TP 2] has been collected). Additional patients may be enrolled to allow for at least 30 evaluable patients

ELIGIBILITY:
For inclusion in the study patients should fulfil the following criteria:

1. Male or female, aged at least 18 years.
2. Able to eat a high-fat meal within a 30-minute period, as provided by the study site.
3. Histologically or, where appropriate, cytologically confirmed NSCLC.
4. Radiological documentation of disease progression while on a previous continuous treatment with an EGFR TKI. In addition, other lines of therapy may have been given. All patients must have documented radiological progression on the last treatment administered prior to enrolling in the study.
5. Confirmation that the tumour harbours an EGFR mutation known to be associated with EGFR TKI sensitivity (including G719X, exon 19 deletion, L858R, L861Q).
6. ECOG performance status 0-1 with no deterioration over the previous 2 weeks.
7. Patients must have a life expectancy of ≥12 weeks, as estimated at the time of screening.
8. Females should be using adequate contraceptive measures and must have a negative pregnancy test prior to start of dosing if of child-bearing potential, or must have evidence of non-child-bearing potential by fulfilling one of the following criteria at screening: Post-menopausal defined as aged more than 50 years and amenorrhoeic for at least 12 months following cessation of all exogenous hormonal treatments; Women under 50 years old would be considered post-menopausal if they have been amenorrhoeic for 12 months or more following cessation of exogenous hormonal treatments and with luteinizing hormone and follicle stimulating hormone levels in the post-menopausal range for the institution; Documentation of irreversible surgical sterilisation by hysterectomy, bilateral oophorectomy, or bilateral salpingectomy, but not tubal ligation.
9. Male patients should be willing to use barrier contraception, ie, condoms, until 6 months after last study drug is taken.

Patients should not enter the study if any of the following exclusion criteria are fulfilled:

1. Participation in another clinical study with an IP during the last 14 days (or a longer period depending on the defined characteristics of the agents used).
2. Treatment with any of the following: Treatment with an EGFR TKI w/in 8 days or approximately 5x half-life, whichever is the longer, of the first dose of study treatment; Any cytotoxic chemotherapy, investigational agents or other anticancer drugs w/in 14 days of the first dose of study treatment; Major surgery (excluding placement of vascular access) within 4 weeks of the first dose; Radiotherapy with a limited field of radiation for palliation within 1 week of the first dose of study treatment, with the exception of patients receiving radiation to more than 30% of the bone marrow or with a wide field of radiation which must be completed within 4 weeks of the first dose of study treatment; Patients currently receiving (or unable to stop use prior to receiving the first dose of study treatment) medications or herbal supplements known to be potent inhibitors of CYP2C8 and of CYP3A4 (at least 1 week prior) and potent inducers of CYP3A4 (at least 3 week prior). All patients must try to avoid concomitant use of any medications, herbal supplements and/or ingestion of foods with known inducer/inhibitory effects on CYP3A4, CYP2C8, and/ or CYP1A2.
3. Any intake of grapefruit, grapefruit juice, Seville oranges, Seville orange marmalade, or other products containing grapefruit or Seville oranges within 7 days of the first administration of the IP until the end of Part A.
4. Any unresolved toxicities from prior therapy greater than CTCAE Grade 1 at the time of starting study treatment with the exception of alopecia and Grade 2, prior platinum therapy related neuropathy.
5. Patients unable to fast for up to 14 hours.
6. Spinal cord compression or brain metastases unless asymptomatic, stable and not requiring steroids for at least 4 weeks prior to start of study treatment.
7. Any evidence of severe or uncontrolled systemic diseases, including uncontrolled hypertension and active bleeding diatheses, which in the Investigator's opinion makes it undesirable for the patient to participate in the study or which would jeopardise compliance with the protocol, or active infection including hepatitis B, hepatitis C and human immunodeficiency virus. Screening for chronic conditions is not required.
8. Patients with type I diabetes.
9. Patients unable to swallow orally administered medication or patients with gastrointestinal disorders or significant gastrointestinal resection likely to interfere with the absorption of AZD9291.
10. Past medical history of ILD, drug-induced ILD, radiation pneumonitis which required steroid treatment, or any evidence of clinically active ILD.
11. Women who are breastfeeding.
12. Patients with a known hypersensitivity to AZD9291
13. Inadequate bone marrow reserve or organ function as demonstrated by any of the following laboratory values: Absolute neutrophil count (ANC) <1.5 x 109/L; Platelet count <100 x 109/L; Haemoglobin <90 g/L; ALT >2.5 x the institutional ULN if no demonstrable liver metastases or >5 x institutional ULN in the presence of liver metastases; AST >2.5 x institutional ULN if no demonstrable liver metastases or >5 x institutional ULN in the presence of liver metastases; Total bilirubin >1.5 x institutional ULN if no liver metastases or >3 x institutional ULN in the presence of documented Gilbert's Syndrome (unconjugated hyperbilirubinaemia) or liver metastases; Creatinine >1.5 x institutional ULN concurrent with creatinine clearance <50 mL/min (measured or calculated by Cockcroft-Gault formula); confirmation of creatinine clearance is only required when creatinine is >1.5 x institutional ULN.
14. Any of the following cardiac criteria: Mean resting corrected QT interval corrected for heart rate using Fridericia's correction factor (QTcF) >470 msec obtained from 3 ECGs; Any clinically important abnormalities in rhythm, conduction or morphology of resting ECG eg, complete left bundle branch block, third degree heart block, second degree heart block, PR interval >250 msec; Any factors that increase the risk of QTc prolongation or risk of arrhythmic events such as heart failure, hypokalaemia, congenital long QT syndrome, family history of long QT syndrome or unexplained sudden death under 40 years of age or any concomitant medication known to prolong the QT interval.
15. For optional genetic research: Previous allogenic bone marrow transplant or non-leukocyte depleted whole blood transfusion within 120 days of the date of the genetic sample collection.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2014-11-14 (Actual); Primary Completion 2015-03-24 (Actual); Study Completion 2023-01-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Serban Ghiorghiu, MSD, Study Director — AstraZeneca
Locations (10):
- France (3):
  - Research Site, Dijon
  - Research Site, Lyon
  - Research Site, Saint-Herblain
- Research Site, Seoul, South Korea
- Spain (2):
  - Research Site, Madrid
  - Research Site, Seville
- United Kingdom (4):
  - Research Site, London
  - Research Site, Manchester
  - Research Site, Newcastle upon Tyne
  - Research Site, Sutton

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] Vishwanathan K, Dickinson PA, Bui K, Cassier PA, Greystoke A, Lisbon E, Moreno V, So K, Thomas K, Weilert D, Yap TA, Plummer R. The Effect of Food or Omeprazole on the Pharmacokinetics of Osimertinib in Patients With Non-Small-Cell Lung Cancer and in Healthy Volunteers. J Clin Pharmacol. 2018 Apr;58(4):474-484. doi: 10.1002/jcph.1035. Epub 2017 Nov 26. PMID 29178442
- See also: Study9_Redacted — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=2987&filename=Study9_Redacted.pdf
- See also: CSR Synopsis Redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D5160C00009&attachmentIdentifier=4f5d7dd7-6acc-4e98-8414-3323c1167aca&fileName=CSR_Synopsis_Redacted.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First subject enrolled: 14 November 2014; Last Subject Last Visit for Part A: 23 March 2015 and Part B: 22 March 2016. The study was performed at 12 sites across Asia and Western Europe. Part A determined effect of food on PK of AZD9291; Part B allowed subjects further access to AZD9291 and provided additional safety data.
Pre-assignment Details: 43 subjects were enrolled (signed informed consent). Subjects were assigned to treatment if they met all the inclusion and none of the exclusion criteria. 5 subjects were enrolled but failed inclusion/exclusion criteria and so were not eligible to be assigned treatment. The remaining 38 subjects started Period 1 and received treatment.
Groups:
- Fed/Fasted: In Part A of the study, each patient received a single 80 mg oral AZD9291 tablet dose in each of 2 treatment periods. Patients who were randomised to the Fed/Fasted treatment group followed Sequence 1: AZD9291 tablets following a high-fat meal in Period 1, then AZD9291 tablets following a period of fasting in Period 2.
- Fasted/Fed: In Part A of the study, each patient received a single 80 mg oral AZD9291 tablet dose in each of 2 treatment periods. Patients who were randomised to the Fasted/Fed treatment group followed Sequence 2: AZD9291 tablets following a period of fasting in Period 1, then AZD9291 tablets following a high-fat meal in Period 2.
- AZD9291 Alone (Part B): In Part B of the study, each patient (who completed Part A) received 80 mg oral AZD9291 tablet formulation once daily, for the duration of their participation.
Period: Part A: Day 1-9 (1st Intervention)
Arm/Group | Fed/Fasted | Fasted/Fed | AZD9291 Alone (Part B)
Started | 18 | 20 | 0
Completed | 18 | 20 | 0
Not Completed | 0 | 0 | 0
Period: Part A: Day 10-15 (2nd Intervention)
Arm/Group | Fed/Fasted | Fasted/Fed | AZD9291 Alone (Part B)
Started | 18 | 20 | 0
Completed | 18 | 20 | 0
Not Completed | 0 | 0 | 0
Period: Part B: Day 15 to End Part B (AZD9291)
Arm/Group | Fed/Fasted | Fasted/Fed | AZD9291 Alone (Part B)
Started | 0 (Only the AZD9291 once daily (Part B) arm is applicable for this period.) | 0 (Only the AZD9291 once daily (Part B) arm is applicable for this period.) | 38 (No patients completed previous period as relates to Part A and arm is applicable only for Part B.)
Completed | 0 | 0 | 14
Not Completed | 0 | 0 | 24
Not completed — Death | 0 | 0 | 5
Not completed — Disease progression | 0 | 0 | 19

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fed/Fasted | Fasted/Fed | Total
Number analyzed (Participants) | 18 | 20 | 38
Age, Continuous [Mean (Standard Deviation); unit: Years] | 64.1 (11.98) | 61.4 (11.00) | 62.7 (11.40)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 10 | 26
  Male | 2 | 10 | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 4 | 2 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 14 | 17 | 31
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: AUC(0-72) of AZD9291
Description: Pharmacokinetics of AZD9291 by assessment of area under the plasma concentration time curve from zero to 72 hours.
Time Frame: Blood samples collected on Day 1 and Day 10 at pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 48 and 72 hours post AZD9291 dose in Part A.
Population: All patients who received at least 1 dose of AZD9291 and had sufficient postdose PK assessments to determine parameter without important protocol deviations/violations and excluding Period 2 data for patients meeting carry-over exclusion criterion (defined as Period 2 pre-dose concentration >5% of Cmax).
Measure: Geometric Mean (Full Range); unit: nM*h
Groups:
- Fed (High-fat Meal): AZD9291 tablets following a high-fat meal
Arm/Group | Fed (High-fat Meal) | Fasted
Number analyzed (Participants) | 26 | 22
nM*h | 7403 [3170 to 15600] | 7345 [3400 to 14700]
Statistical Analysis 1: Comparison: Fed (High-fat Meal) vs Fasted; Study sized so experiment-wise power for the 90% CIs of geometric mean ratios for both AUC and Cmax of AZD9291 being within 70-143% was 90% (95% for each parameter). Within patient CV assumed to be 34%. A 6% change in exposure was also assumed; Test type: Non-Inferiority or Equivalence — 90% CIs being within 70% to 143%; Geometric mean ratio = 106.05, 90% CI 2-sided [94.82 to 118.60] — Fed / Fasted ratio. Linear mixed-effects model with sequence, period, and treatment as fixed effects and subject nested within sequence as a random effect. Least squares geometric mean ratio (LSGMR) Fed = 7847, Fasted = 7399

2. Primary Outcome: Cmax of AZD9291
Description: Pharmacokinetics of AZD9291 by assessment of maximum plasma AZD9291 concentration.
Time Frame: Blood samples collected on Day 1 and Day 10 at pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72, 120, 168, and 216 hours post AZD9291 dose in Part A.
Population: All patients had at least 1 dose AZD9291 and had sufficient postdose PK to determine parameter without important protocol deviations and excluding Period 2 data for patients meeting carry-over exclusion criterion (defined as Period 2 pre-dose concentration >5% of Cmax). Note 1 patient missing key 8 hour sample so not included in Cmax analysis.
Measure: Geometric Mean (Full Range); unit: nM
Arm/Group | Fed (High-fat Meal) | Fasted
Number analyzed (Participants) | 25 | 22
nM | 199.6 [80.8 to 446] | 218.0 [95.2 to 381]
Statistical Analysis 1: Comparison: Fed (High-fat Meal) vs Fasted; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — 90% CIs being within 70% to 143%; Geometric mean ratio = 92.75, 90% CI 2-sided [81.40 to 105.68] — Fed / Fasted ratio. Linear mixed-effects model with sequence, period, and treatment as fixed effects and subject nested within sequence as a random effect. LSGMR Fed = 208.0, Fasted = 224.3

3. Secondary Outcome: AUC of AZD9291
Description: Area under the plasma concentration curve from zero extrapolated to infinity.
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Geometric Mean (Full Range); unit: nM*h
Arm/Group | Fed (High-fat Meal) | Fasted
Number analyzed (Participants) | 22 | 19
nM*h | 11640 [5460 to 24100] | 12530 [6050 to 25500]

4. Secondary Outcome: AUC(0-t) of AZD9291
Description: Area under the plasma concentration curve from time zero to last quantifiable dose.
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Geometric Mean (Full Range); unit: nM*h
Arm/Group | Fed (High-fat Meal) | Fasted
Number analyzed (Participants) | 26 | 22
nM*h | 10820 [4860 to 21800] | 10630 [5300 to 22600]

5. Secondary Outcome: AUC(0-120) of AZD9291
Description: Pharmacokinetics of AZD9291 by assessment of area under the plasma concentration time curve from zero to 120 hours.
Time Frame: Blood samples collected on Day 1 and Day 10 at pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72 and 120 hours post AZD9291 dose in Part A.
Population: as for outcome 1
Measure: Geometric Mean (Full Range); unit: nM*h
Arm/Group | Fed (High-fat Meal) | Fasted
Number analyzed (Participants) | 25 | 21
nM*h | 9549 [4360 to 18800] | 9308 [4480 to 18900]

6. Secondary Outcome: Tmax of AZD9291
Description: Pharmacokinetics of AZD9291 by assessment of time to Cmax.
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Median (Full Range); unit: h
Arm/Group | Fed (High-fat Meal) | Fasted
Number analyzed (Participants) | 25 | 22
h | 7.97 [3.02 to 24.13] | 6.08 [3.00 to 10.07]

7. Secondary Outcome: t1/2 of AZD9291
Description: Pharmacokinetics of AZD9291 by assessment of the terminal half-life.
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Geometric Mean (Full Range); unit: h
Arm/Group | Fed (High-fat Meal) | Fasted
Number analyzed (Participants) | 25 | 21
h | 52.82 [32.1 to 84.4] | 54.64 [31.2 to 84.0]

8. Secondary Outcome: CL/F of AZD9291
Description: Rate and extent of absorption of AZD9291 by assessment of apparent clearance following oral administration.
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Geometric Mean (Full Range); unit: L/h
Arm/Group | Fed (High-fat Meal) | Fasted
Number analyzed (Participants) | 22 | 19
L/h | 13.75 [6.65 to 29.3] | 12.78 [6.28 to 26.5]

9. Secondary Outcome: Vz/F of AZD9291
Description: Rate and extent of absorption of AZD9291 by assessment of the apprarent volume of distribution.
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Geometric Mean (Full Range); unit: L
Arm/Group | Fed (High-fat Meal) | Fasted
Number analyzed (Participants) | 22 | 19
L | 1024 [470 to 2580] | 1019 [432 to 2200]

10. Secondary Outcome: AUC(0-72) of AZ5104 and AZ7550
Description: Pharmacokinetics of AZ5104 and AZ7550 (metabolites to AZD9291) by assessment of area under the plasma concentration time curve from zero to 72 hours.
Time Frame: as for outcome 1
Population: All patients who received at least 1 dose of AZD9291 and had sufficient postdose PK assessments to determine parameter without important protocol deviations/violations and excluding Period 2 data for patients meeting carry-over exclusion criterion (defined as Period 2 pre-dose concentration >10% of Cmax for respective metabolite).
Measure: Geometric Mean (Full Range); unit: nM*h
Arm/Group | Fed (High-fat Meal) | Fasted
Number analyzed (Participants) | 17 | 17
nM*h
  AZ5104 | 497.6 [138 to 1360] | 613.2 [270 to 1450]
  AZ7550 | 235.0 [82.7 to 1140] | 266.4 [112 to 590]
Statistical Analysis 1: Comparison: Fed (High-fat Meal) vs Fasted; AZ5104; Test type: Superiority or Other; Geometric mean ratio = 81.15, 90% CI 2-sided [57.86 to 113.83] — Fed / Fasted ratio. No pre-specified margins for equivalence test for metabolites, but analysed for consistency with AZD9291 analysis. Linear mixed-effects model with treatment as fixed effect. LSGMR Fed = 497.6, Fasted = 613.2
Statistical Analysis 2: Comparison: Fed (High-fat Meal) vs Fasted; AZ7550; Test type: Superiority or Other; Geometric mean ratio = 88.21, 90% CI 2-sided [65.21 to 119.32] — Fed / Fasted ratio. No pre-specified margins for equivalence test for metabolites, but analysed for consistency with AZD9291 analysis. Linear mixed-effects model with treatment as fixed effect. LSGMR Fed = 235.0, Fasted = 266.4

11. Secondary Outcome: Cmax of AZ5104 and AZ7550
Description: Pharmacokinetics of AZ5104 and AZ7550 (metabolites to AZD9291) by assessment of maximum plasma concentration.
Time Frame: as for outcome 2
Population: as for outcome 10
Measure: Geometric Mean (Full Range); unit: nM
Arm/Group | Fed (High-fat Meal) | Fasted
Number analyzed (Participants) | 17 | 17
nM
  AZ5104 | 9.163 [2.94 to 24.7] | 11.95 [4.95 to 28.6]
  AZ7550 | 4.236 [1.76 to 19.7] | 5.109 [1.78 to 11.3]
Statistical Analysis 1: Comparison: Fed (High-fat Meal) vs Fasted; AZ5104; Test type: Superiority or Other; Geometric mean ratio = 76.68, 90% CI 2-sided [55.31 to 106.32] — Fed / Fasted ratio. No pre-specified margins for equivalence test for metabolites, but analysed for consistency with AZD9291 analysis. Linear mixed-effects model with treatment as fixed effect. LSGMR Fed = 9.163, Fasted = 11.95
Statistical Analysis 2: Comparison: Fed (High-fat Meal) vs Fasted; AZ7550; Test type: Superiority or Other; Geometric mean ratio = 82.92, 90% CI 2-sided [60.99 to 112.74] — Fed / Fasted ratio. No pre-specified margins for equivalence test for metabolites, but analysed for consistency with AZD9291 analysis. Linear mixed-effects model with treatment as fixed effect. LSGMR Fed = 4.236, Fasted = 5.109

12. Secondary Outcome: AUC(0-t) of AZ5104 and AZ7550
Description: Area under the plasma concentration curve from time zero to last quantifiable dose for AZ5104 and AZ7550 (metabolites to AZD9291).
Time Frame: as for outcome 2
Population: as for outcome 10
Measure: Geometric Mean (Full Range); unit: nM*h
Arm/Group | Fed (High-fat Meal) | Fasted
Number analyzed (Participants) | 17 | 17
nM*h
  AZ5104 | 1033 [266 to 2590] | 1132 [535 to 2640]
  AZ7550 | 584.5 [178 to 2530] | 591.9 [270 to 1090]

13. Secondary Outcome: AUC(0-120) of AZ5104 and AZ7550
Description: Pharmacokinetics of AZ5104 and AZ7550 (metabolites to AZD9291) by assessment of area under the plasma concentration time curve from zero to 120 hours.
Time Frame: as for outcome 5
Population: as for outcome 10
Measure: Geometric Mean (Full Range); unit: nM*h
Arm/Group | Fed (High-fat Meal) | Fasted
Number analyzed (Participants) | 16 | 17
nM*h
  AZ5104 | 744.4 [206 to 2050] | 875.7 [408 to 1940]
  AZ7550 | 373.4 [127 to 1820] | 411.4 [178 to 850]

14. Secondary Outcome: Tmax of AZ5104 and AZ7550
Description: Pharmacokinetics of AZ5104 and AZ7550 (metabolites to AZD9291) by assessment of time to Cmax.
Time Frame: as for outcome 2
Population: as for outcome 10
Measure: Median (Full Range); unit: h
Arm/Group | Fed (High-fat Meal) | Fasted
Number analyzed (Participants) | 17 | 17
h
  AZ5104 | 24.17 [8.08 to 72.75] | 8.03 [4.00 to 49.03]
  AZ7550 | 24.60 [8.08 to 120.58] | 10.00 [6.00 to 73.53]

15. Secondary Outcome: t1/2 of AZ5104 and AZ7550
Description: Pharmacokinetics of AZ5104 and AZ7550 (metabolites to AZD9291) by assessment of the terminal half-life.
Time Frame: as for outcome 2
Population: as for outcome 10
Measure: Geometric Mean (Full Range); unit: h
Arm/Group | Fed (High-fat Meal) | Fasted
Number analyzed (Participants) | 17 | 17
h
  AZ5104 | 64.74 [45.9 to 113] | 62.89 [43.3 to 96.2]
  AZ7550 | 85.26 [52.2 to 142] | 91.54 [58.2 to 204]

ADVERSE EVENTS:
Time Frame: Approximately 2 weeks for Part A; up to approximately 15 months for Part B and approximately 15.5 months for Overall (Parts A and B combined).
Description: Part A: Adverse events (AEs) collected from day of first dose until day prior to first dose in Part B (Day 15), or until 30 days after last dose if discontinued in Part A. Part B: AEs collected from day of first dose in Part B until 30 days after last dose, or until last dose in Part B for those entering continued access phase (CAP).
Groups:
- Overall Safety Population: Parts A and B of the study combined.
- Part A Safety Population: In Part A of the study, each patient received a single 80 mg oral AZD9291 tablet dose in each of 2 treatment periods. Patients were randomised to either Sequence 1 (AZD9291 tablets following a high-fat meal in Period 1, then AZD9291 tablets following a period of fasting in Period 2) or Sequence 2 (AZD9291 tablets following a period of fasting in Period 1, then AZD9291 tablets following a high-fat meal in Period 2).
- Part B Safety Population: In Part B of the study, each patient received 80 mg oral AZD9291 tablet formulation once daily, for the duration of their participation.
Arm/Group | Overall Safety Population | Part A Safety Population | Part B Safety Population
All-Cause Mortality (participants affected / at risk) | 2/38 | 0/38 | 2/38
Serious Adverse Events (participants affected / at risk) | 8/38 | 1/38 | 7/38
Other Adverse Events (participants affected / at risk) | 38/38 | 20/38 | 37/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Overall Safety Population (N=38) | Part A Safety Population (N=38) | Part B Safety Population (N=38)
ATRIAL FLUTTER (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
LOWER RESPIRATORY TRACT INFECTION BACTERIAL (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
NEUTROPENIC SEPSIS (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
PNEUMONIA (Infections and infestations) | 2 (2) | 0 (0) | 2 (2) — Death in 1 subject (same subject as Sepsis fatal outcome SAE)
PNEUMONIA PNEUMOCOCCAL (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
SEPSIS (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) — Death (same subject as Pneumonia fatal outcome SAE)
HYPONATRAEMIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
INTERVERTEBRAL DISC COMPRESSION (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
CANCER PAIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1)
HEADACHE (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
RESPIRATORY DISTRESS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) — Death
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Overall Safety Population (N=38) | Part A Safety Population (N=38) | Part B Safety Population (N=38)
ANAEMIA (Blood and lymphatic system disorders) | 6 (6) | 3 (3) | 3 (3)
NEUTROPENIA (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 2 (2)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 4 (4) | 1 (1) | 3 (3)
BLEPHARITIS (Eye disorders) | 2 (2) | 0 (0) | 2 (2)
CATARACT (Eye disorders) | 3 (3) | 0 (0) | 3 (3)
DRY EYE (Eye disorders) | 5 (5) | 0 (0) | 5 (5)
LACRIMATION INCREASED (Eye disorders) | 3 (3) | 0 (0) | 3 (3)
VISUAL ACUITY REDUCED (Eye disorders) | 2 (2) | 0 (0) | 2 (2)
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 2 (2) | 0 (0) | 2 (2)
ABDOMINAL PAIN (Gastrointestinal disorders) | 3 (3) | 0 (0) | 3 (3)
CONSTIPATION (Gastrointestinal disorders) | 4 (4) | 0 (0) | 4 (4)
DENTAL CARIES (Gastrointestinal disorders) | 2 (2) | 0 (0) | 2 (2)
DIARRHOEA (Gastrointestinal disorders) | 21 (45) | 4 (4) | 19 (41)
DRY MOUTH (Gastrointestinal disorders) | 2 (2) | 0 (0) | 2 (2)
DYSPEPSIA (Gastrointestinal disorders) | 2 (2) | 0 (0) | 2 (2)
GASTRITIS (Gastrointestinal disorders) | 3 (3) | 0 (0) | 3 (3)
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 3 (3) | 0 (0) | 3 (3)
NAUSEA (Gastrointestinal disorders) | 10 (12) | 4 (4) | 8 (8)
STOMATITIS (Gastrointestinal disorders) | 5 (5) | 0 (0) | 5 (5)
VOMITING (Gastrointestinal disorders) | 6 (17) | 4 (7) | 5 (10)
ASTHENIA (General disorders) | 5 (7) | 1 (1) | 4 (6)
FATIGUE (General disorders) | 9 (10) | 1 (1) | 8 (9)
NON-CARDIAC CHEST PAIN (General disorders) | 2 (2) | 0 (0) | 2 (2)
OEDEMA PERIPHERAL (General disorders) | 4 (5) | 0 (0) | 4 (5)
PYREXIA (General disorders) | 2 (2) | 0 (0) | 2 (2)
BRONCHITIS (Infections and infestations) | 2 (2) | 0 (0) | 2 (2)
CONJUNCTIVITIS (Infections and infestations) | 3 (4) | 1 (1) | 2 (3)
GASTROENTERITIS (Infections and infestations) | 2 (2) | 0 (0) | 2 (2)
LOWER RESPIRATORY TRACT INFECTION (Infections and infestations) | 2 (2) | 0 (0) | 2 (2)
NASOPHARYNGITIS (Infections and infestations) | 2 (3) | 0 (0) | 2 (3)
ORAL CANDIDIASIS (Infections and infestations) | 2 (3) | 1 (1) | 2 (2)
PARONYCHIA (Infections and infestations) | 10 (12) | 1 (1) | 9 (11)
PHARYNGITIS (Infections and infestations) | 2 (2) | 0 (0) | 2 (2)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 4 (5) | 0 (0) | 4 (5)
URINARY TRACT INFECTION (Infections and infestations) | 2 (3) | 0 (0) | 2 (3)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 4 (6) | 0 (0) | 4 (6)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 4 (7) | 0 (0) | 4 (7)
BLOOD CREATININE INCREASED (Investigations) | 2 (2) | 0 (0) | 2 (2)
NEUTROPHIL COUNT DECREASED (Investigations) | 2 (2) | 0 (0) | 2 (2)
WEIGHT DECREASED (Investigations) | 2 (2) | 0 (0) | 2 (2)
DECREASED APPETITE (Metabolism and nutrition disorders) | 10 (12) | 1 (1) | 9 (11)
HYPOKALAEMIA (Metabolism and nutrition disorders) | 3 (4) | 1 (1) | 2 (3)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 5 (5) | 0 (0) | 5 (5)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 8 (8) | 1 (1) | 7 (7)
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 4 (4) | 0 (0) | 4 (4)
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 2 (3) | 0 (0) | 2 (3)
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 6 (7) | 1 (1) | 6 (6)
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 4 (4) | 0 (0) | 4 (4)
BALANCE DISORDER (Nervous system disorders) | 2 (2) | 0 (0) | 2 (2)
DIZZINESS (Nervous system disorders) | 2 (2) | 0 (0) | 2 (2)
HEADACHE (Nervous system disorders) | 6 (11) | 3 (4) | 5 (7)
PARAESTHESIA (Nervous system disorders) | 2 (2) | 0 (0) | 2 (2)
SCIATICA (Nervous system disorders) | 2 (2) | 0 (0) | 2 (2)
SOMNOLENCE (Nervous system disorders) | 2 (2) | 0 (0) | 2 (2)
INSOMNIA (Psychiatric disorders) | 4 (4) | 2 (2) | 2 (2)
POLLAKIURIA (Renal and urinary disorders) | 2 (2) | 0 (0) | 2 (2)
COUGH (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 0 (0) | 6 (6)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 6 (7) | 1 (1) | 5 (6)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 3 (4) | 0 (0)
PRODUCTIVE COUGH (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 2 (2)
DERMATITIS ACNEIFORM (Skin and subcutaneous tissue disorders) | 6 (7) | 0 (0) | 6 (7)
DRY SKIN (Skin and subcutaneous tissue disorders) | 12 (12) | 0 (0) | 12 (12)
NAIL RIDGING (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0) | 3 (3)
PRURITUS (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0) | 3 (3)
RASH (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 2 (2)
RASH ERYTHEMATOUS (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 2 (2)
RASH MACULAR (Skin and subcutaneous tissue disorders) | 5 (5) | 1 (1) | 4 (4)
RASH MACULO-PAPULAR (Skin and subcutaneous tissue disorders) | 4 (4) | 0 (0) | 4 (4)
HYPOTENSION (Vascular disorders) | 2 (2) | 2 (2) | 0 (0)

LIMITATIONS AND CAVEATS:
At end of Part B, the CAP allowed patients to continue receiving AZD9291 if still deriving clinical benefit. No clinical data was databased during the CAP; thus AE data is presented to end of Part B only.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Principal Investigator (PI) agrees to collaborate on the contents and formation of any publication and to pay due consideration to comments and opinions offered. AstraZeneca have 30 days for final manuscript review and may require that submission for publication be delayed in order to file patent application.